CLINICAL TRIAL: NCT01403571
Title: Efficacy and Safety of Whole Grain Salba (Salvia Hispanica L.) on Weight Loss in Overweight and Obese Individuals With Type 2 Diabetes
Brief Title: Effectiveness and Safety of Salba on Weight Loss in Overweight Individuals With Type 2 Diabetes
Acronym: LOSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2103038AJ
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salba supplement (Experimental): 30g/1000kal
  Interventions: Dietary Supplement: Salba (Salvia hispanica L.)
- Oat-bran based Control Supplement (Placebo Comparator): 36g/1000kcal
  Interventions: Dietary Supplement: Oat-based Control

INTERVENTIONS:
Dietary Supplement: Salba (Salvia hispanica L.) — 30g/1000kcal/day over 24 wks
  Arms: Salba supplement
Dietary Supplement: Oat-based Control — Placebo: 36g/1000kcal/day over 24 weeks
  Arms: Oat-bran based Control Supplement

SUMMARY:
Canadian statistics indicate that the incidence of obesity is increasing and that the occurrence of diabetes in obese individuals is 5-fold greater than those with a healthy weight, making weight control in this population particularly relevant. Preliminary clinical data has shown that the whole grain, Salba, may improve type 2 diabetes control, reduce after-meal blood glucose, cardiovascular disease (CVD) risk factors and suppress appetite. Its use may therefore have potential implications in long-term weight management, while improving diabetes.

The objective of this research (weight loss) is to evaluate whether adding Salba to an energy reduced diet for six months will result in greater weight loss compared to control in overweight and obese individuals with type 2 diabetes. The study recruited 77 overweight or obese individuals with type 2 diabetes. They were instructed to follow a calorie restricted diet and their regular diabetes therapy together with regular exercise. Participants were randomly assigned to receive 30 g Salba/1000 kcal of daily energy requirements, or an oat bran control supplement matched for energy. The effect of the supplements on weight-loss (including waist circumference, % body fat) and glucose control (A1c, fasting glucose levels) will be assessed. In addition, related outcomes such as low-grade body inflammation, hunger-regulating hormones (ghrelin, adiponectin), safety measures (urea, creatinine, ALT and prothrombin time) and satiety scores were evaluated.

Modest weight loss has been associated with improved glucose control in individuals with type 2 diabetes. Addition of Salba to an energy reduced diet may facilitate greater weight loss and improve glycemic control and CVD risk factors compared to such a diet alone. Salba may also promote maintenance of weight loss and therefore help prevent weight gain by providing feelings of fullness that reduce appetite. In light of the high incidence of obesity in individuals with diabetes, Salba grain may be a useful addition to the diet.

ELIGIBILITY:
Inclusion Criteria:

* Well-controlled type 2 diabetes for at least 1 year
* Treated with diet and/or oral hypoglycemic medications
* BMI 25-40 kg/m2

Exclusion Criteria:

* Weight change in the past three months >10% of body weight
* On insulin therapy
* Unstable angina, myocardial infarction or stroke (within 6 months)
* Planned surgery or pregnancy
* Blood pressure >160mmHg/100mmHg
* Surgical procedures for weight loss and concomitant use of medication or supplements that alter body weight or appetite
* ALA, dietary fibre, fish oil supplements or consuming cold-water fish more than three times per week

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Weight | 24 weeks
  24 week timeframe for Weightloss phase

SECONDARY OUTCOMES:
Body composition | 24 weeks
  24 week timeframe for Weightloss phase
Blood sugar control | 24 weeks
  (HbA1c and Fasting glucose) 24 week timeframe for Weightloss phase
Low grade body inflammation | 24 weeks
  hs-CRP levels
serum ALT | 24 weeks
  Safety Measures
Prothrombin time | 24 weeks
  Safety Measures
serum creatinine | 24 weeks
  Safety Measures
Blood urea | 24 weeks
  Safety Measures
Satiety hormones | 24 weeks
  ghrelin, adiponectin
Fatty Acids (% composition) | 24 weeks
  ALA (18:3 n-3), LA (18:2 n-6); Compliance measure

CONTACTS AND LOCATIONS:
Locations (1):
- Risk Factor Modification Centre, St. Michael's, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vuksan V, Jenkins AL, Brissette C, Choleva L, Jovanovski E, Gibbs AL, Bazinet RP, Au-Yeung F, Zurbau A, Ho HV, Duvnjak L, Sievenpiper JL, Josse RG, Hanna A. Salba-chia (Salvia hispanica L.) in the treatment of overweight and obese patients with type 2 diabetes: A double-blind randomized controlled trial. Nutr Metab Cardiovasc Dis. 2017 Feb;27(2):138-146. doi: 10.1016/j.numecd.2016.11.124. Epub 2016 Dec 9. PMID 28089080